CLINICAL TRIAL: NCT04854824
Title: A Simple, Home-treatment Algorithm to Prevent Hospitalization for COVID-19 Patients: A Matched -Cohort Study
Brief Title: A Simple Approach to Prevent Hospitalization for COVID-19 Patients
Acronym: COVER2
Status: Completed | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: COVER 2
Record Dates: First submitted 2021-04-21; First posted 2021-04-22 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Covid19
Keywords: COVID-19 treatment at home; Early symptoms; Hospitalization
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 'Recommended algorithm' cohort: COVID-19 patients treated at home by their family doctors according to the proposed recommendations
  Interventions: Drug: Recommended treatment schedule
- 'Historic control' cohort: COVID-19 patients enrolled in the ORIGIN study of the Istituto di Ricerche Farmacologiche Mario Negri IRCCS and treated at home by family physicians with drug regimens that are not necessarily guided by those proposed in the recommendations
  Interventions: Drug: Control treatment schedule

INTERVENTIONS:
Drug: Recommended treatment schedule — Relatively selective Cox-2 inhibitors, Corticosteroids (Dexamethasone), Anticoagulants (LMW heparin), Gentle oxygen therapy
  Groups: 'Recommended algorithm' cohort
Drug: Control treatment schedule — Treatment regimens different from the recommended one according to family physician personal practice
  Groups: 'Historic control' cohort

SUMMARY:
The newly recognised disease COVID-19 is caused by the Severe-Acute-Respiratory-Syndrome Coronavirus 2 (SARS-CoV-2), which rapidly spread globally in late 2019, reaching pandemic proportions. The clinical spectrum of SARS-CoV-2 infection is broad, encompassing asymptomatic infection, mild upper respiratory tract illness and mild extrapulmonary symptoms, and severe viral pneumonia with respiratory failure and even death.

Given the rising global death toll associated with the pandemic, in the last year we have witnessed a race to find drugs/biological treatments to save the lives of hospitalised, severely ill patients, as well as to develop vaccines. Nonetheless, to limit the number of hospitalisations and deaths due to severe illness, thus avoiding pushing hospitals to their limits and remarkably reducing the tremendous treatment costs for health care providers, it is crucial to also focus on primary care physicians and initial mild symptoms in COVID-19 patients at home.

As with other acute viral infections, early initiation of treatment for COVID-19 might improve clinical outcomes.

For COVID-19, most primary care physicians have initially treated their patients according to their judgment, with various treatment regimens they believe are most appropriate based on thier experience/expertise. We recently published a note on how we were treating patients at home based on the pathophysiologic and pharmacologic rationale and the available clinical evidence of efficacy in COVID-19 for each of the recommended class of drugs.

Because the common early mild symptoms of COVID-19 highlight a systemic inflammatory process, there is the recommendation of using anti-inflammatory agents to limit excessive host inflammatory responses to the viral infection, including non-steroidal anti-inflammatory drugs and corticosteroids.

In a recent academic matched-cohort study, we found that early treatment of COVID-19 patients at home by their family doctors according to the proposed recommendation regimen almost completely prevented the need for hospital admission (the most clinically relevant outcome) due to progression toward more severe illness, compared to patients in the 'control' cohort who were treated at home according to their family physician's assessments. This translated into a reduction of over 90% in the overall numbers of days of hospitalisation and in related treatment costs. Treatment according to the recommended algorithm was safe and well tolerated. However, the rate of hospitalization was a secondary outcome of the study and the possibility of a casual finding cannot be definitely excluded. Thus, we have considered the observed reduction in patient hospitalization an hypothesis generating finding that provides a robust background for the present new cohort study primarily aimed to test the effect on this outcome of COVID-19 treatment at home according to the proposed recommendation algorithm.

No randomized clinical trials have been performed so far in COVID-19 patients to compare the effectiveness of different regimens targeting early symptoms at home. Comparative analysis of patient cohorts with long-enough follow-up in everyday clinical practice may offer a good alternative to randomized clinical trials to evaluate effectiveness of therapeutic interventions. Thus, we will use this approach to compare a cohort of COVID-19 patients treated at home by their family physicians according to the proposed recommendation algorithm with another cohort of similar COVID-19 patients treated by their family doctors with various treatment regimens they believe most appropriate based on their experience and expertise, and monitored longitudinally up to 3 months.

Our working hypothesis is that following the proposed recommendation algorithm the early COVID-19-related inflammatory process is limited, preventing the need of hospital admission at larger extent than with other therapeutic approaches also targeting early symptoms of the illness at home.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult (≥18 years old)
* Subjects with early mild symptoms of COVID-19, who start the treatment without waiting results of a nasopharyngeal swab, if any
* Informed consent

Exclusion Criteria:

* Subjects of the two cohorts who require immediate hospital admission because of severe COVID-19 symptoms at onset according to family doctor's assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: "Recommended algorithm" cohort COVID-19 patients treated at home by their family doctors according to the proposed recommendations from 1 January 2021 to 30 April 2021. It will include all available family physicians in the Bergamo, Varese and Teramo provinces who have followed the recommendation algorithm and expressed interest in participating in the study.
  "Historic control" cohort Historic COVID-19 patients enrolled in the ORIGIN study, treated at home by their family physicians with drug regimens not necessarily guided by those proposed in the recommendations.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who require hospitalization | From beginning the proposed recommended treatments or other therapeutic regimens, assessed up to 60 days.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - ASL Teramo, Teramo, TE
  - ATS Insubria, Varese, VA

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Consolaro E, Suter F, Rubis N, Pedroni S, Moroni C, Pasto E, Paganini MV, Pravettoni G, Cantarelli U, Perico N, Perna A, Peracchi T, Ruggenenti P, Remuzzi G. A Home-Treatment Algorithm Based on Anti-inflammatory Drugs to Prevent Hospitalization of Patients With Early COVID-19: A Matched-Cohort Study (COVER 2). Front Med (Lausanne). 2022 Apr 22;9:785785. doi: 10.3389/fmed.2022.785785. eCollection 2022. PMID 35530041